CLINICAL TRIAL: NCT06271291
Title: Pancreatic Cancer Detection Consortium (PCDC) Prospective Cohorts
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23-000161; NCI-2024-00504 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-000161 (Other: Mayo Clinic in Rochester); U01CA210138 (NIH); U24CA274496 (NIH)
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens of subjects without pancreatic cancer who are at high-risk for pancreatic cancer due to a strong family history, a mutation in a known pancreatic cancer predisposition gene, or Fukuoka worrisome or high-risk pancreatic cysts. Biospecimens will remain available for research beyond the end of study funding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Participants undergo blood sample collection, complete questionnaires, have their medical records reviewed and undergo pancreatic cyst fluid collection during standard of care endoscopic ultrasounds fine needle aspiration.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates individuals without pancreatic cancer, but who have been determined to be at higher-than-average lifetime risk of developing pancreatic cancer to help detect pancreatic cancer or other cancers at an earlier time when they might be more easily treated and cured.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a cohort (biobank of biospecimens and data) of subjects without pancreatic cancer who are at highrisk for pancreatic cancer due to: a strong family history, a mutation in a known pancreatic cancer predisposition gene, or fukuoka worrisome or high-risk pancreatic cysts.

II. To follow the cohort subjects longitudinally and collect biospecimens and follow-up data and record medical outcomes.

III. To make biospecimen available to PCDC-approved projects to validate potential biomarkers for performance using nested case-control prospective designs.

OUTLINE: This is an observational study.

Participants undergo blood sample collection, complete questionnaires, have their medical records reviewed and undergo pancreatic cyst fluid collection during standard of care endoscopic ultrasounds fine needle aspiration.

ELIGIBILITY:
Inclusion Criteria:

* PDAC FAMILY HISTORY OR PDAC RELATED GENETIC MUTATIONS:

  * Age: 50 or older, plus at least one of the following:

    * Mutation unknown or absent:

      * 2+ relatives with PDAC on same side of family where 2 affected are first degree related to each other and at least 1 affected is first degree related to subject;
      * OR 2+ affected first degree relatives (FDR), defined as blood related parents, siblings, or children)
    * Known pathogenic/likely pathogenic (P/LP) mutation in at least one of the following:

      * CDKN2A/p16, PJS (STK11), Hereditary pancreatitis with confirmed protease serine 1 (PRSS1)
    * OR 1+FDR or second degree relative (SDR) with PDAC and a known P/LP mutation in one or more of:

      * ATM, BRCA1, BRCA2, PALB2, Lynch syndrome (MLH1, MSH2, MSH6, PMS2, EPCAM), TP53

HIGH-RISK OR WORRISOME PANCREATIC CYSTS:

* 18 years of age or greater and meeting Fukuoka worrisome (FW) or Fukuoka high-risk (FHR) criteria

  * High risk stigmata:

    * Obstructive Jaundice in a patient with cystic lesion of the head of the pancreas
    * Enhancing mural nodule ≥ 5 mm
    * Main pancreatic duct ≥ 10 mm
  * Worrisome features:

    * Presence of pancreatic duct stricture, defined as focal pancreatic duct narrowing with upstream duct => 6 mm
    * Cyst ≥ 3 cm
    * Enhancing mural nodule < 5 mm
    * Thickened/Enhancing cyst wall
    * Main duct size 5-9 mm
    * Pancreatitis
    * Lymphadenopathy
    * Increased CA 19-9
    * Cyst growth rate ≥ 5 mm /2 years

Exclusion Criteria:

* * Is unable to provide informed consent

  * Has received a non-autologous bone marrow transplant or has an active hematologic malignancy (i.e., leukemia or lymphoma)
  * Current or prior history of PDAC or total pancreatectomy
  * Is currently a prison inmate
  * Is not able to speak or read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic ductal adenocarcinoma (PDAC) family history, PDAC related genetic mutations or high risk or worrisome pancreatic cysts
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2029-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Develop a biobank of biospecimens and data of subjects without pancreatic cancer who are at high risk for pancreatic cancer | Baseline (at enrollment)
  Assessed by the number of specimens collected for subjects at right risk for pancreatic cancer due to a strong family history, a mutation in a known pancreatic cancer predisposition gene, or Fukuoka worrisome or high-risk pancreatic cysts.
Follow subjects longitudinally and collect biospecimens and follow-up data and record medical outcomes | Up to study completion, as defined in description
  Participants will be followed until study completion, defined as when one or more of the following occur:
  * Subject has provided a pre-treatment biospecimen after diagnosis with pancreatic ductal adenocarcinoma (PDAC) or it has been determined that collection of a pre-treatment biospecimen sample after PDAC diagnosis is infeasible.
  * Enrollment cyst determined to not be mucinous and thus not worthy of ongoing surveillance.
  * Subject has had a complete pancreatectomy.
  * Subject has died.
  * Study funding has ended

CONTACTS AND LOCATIONS:
Overall Officials: Ann L. Oberg, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (5):
- United States (5):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials